CLINICAL TRIAL: NCT05936008
Title: Investigating Exercise Prescription Parameters on Aerobic Fitness and Vascular Health After Stroke: A Pilot Study
Brief Title: Fitness After Stroke Trial
Acronym: FAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Sandra Billinger, Professor and Vice Chair, Stroke Translational Research, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00147598
Record Dates: First submitted 2023-06-19; First posted 2023-07-07 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Stroke, Ischemic; Stroke Hemorrhagic
Keywords: exercise; cerebrovascular; cardiovascular; walking; aerobic fitness; brain
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The Investigator will use an adaptive randomization design called minimization to ensure balance across groups. Intervention arms include:
  1. Moderate intensity, continuous training exercise
  2. High intensity, interval training exercise
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the participant's intervention group. Participants will not be given detailed information about the exercise groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate intensity, continuous training (MICT) (Active Comparator): After a 5-minute warm-up at 30% peak watts, MICT will consist of continuous exercise for 25 minutes at 55% of peak watts (range: 45%-65%). The average heart rate for each individual session should not exceed 70% (60-70%) of HR maximum to align with current exercise recommendations for stroke. An active cool-down (20% peak workload) at comfortable stepping pace occurs immediately after the intervention.
  Interventions: Behavioral: Exercise MICT
- High intensity, interval exercise (HIIT) (Active Comparator): After the 5-minute warm-up at 30% peak watts, HIIT will consist of repeated 1-minute, high intensity bursts ("on" interval) alternated with 1-minute interval recovery ("off" interval) for 25 minutes. The "on" interval will begin at 70% of peak watts (range: 65%-95%) followed by the "off" interval at 10% of peak watts. The average HR for the "on" intervals will not exceed 85% age predicted maximum (75-85%). There will be 13 minutes of "on" and 12 minutes of "off" interval exercise. An active cool-down (20% peak workload) at comfortable stepping pace occurs immediately after the intervention.
  Interventions: Behavioral: Exercise HIIT

INTERVENTIONS:
Behavioral: Exercise MICT — Standard of care, exercise recommendations for people with stroke
  Other Names: aerobic exercise
  Arms: Moderate intensity, continuous training (MICT)
Behavioral: Exercise HIIT — The HIIT protocol consists of Short Interval, High Volume exercise at 1-minute exercise bouts followed by 1-minute active recovery for 25 minutes.
  Other Names: HIIT, aerobic exercise, anaerobic exercise
  Arms: High intensity, interval exercise (HIIT)

SUMMARY:
People living with stroke have very low aerobic fitness, which can negatively impact brain health. Identifying the best exercise which includes exercise stimulus type (interval, continuous) or intensity, how hard to exercise (moderate, high) that benefit aerobic fitness, vascular health, and the brain's main blood vessels after stroke are unknown. This study is designed to determine the preliminary efficacy of high-volume HIIT to moderate intensity exercise using a seated stepper exercise device that allows the arms and legs to move back and forth.

DETAILED DESCRIPTION:
People with stroke often experience physical decline and aerobic fitness that can be reversed through exercise. Evidence has shown that participating in exercise benefits aerobic fitness and vascular health while less is known about brain health. However, the optimal exercise dose such as intensity and exercise type (continuous, interval) are not yet known.

The long-term goal of this project is to develop and test strategies to be implemented in larger clinical trials to improve health in people living with stroke. For this preliminary efficacy trial, the Investigator will enroll 50 participants with chronic stroke, age 20-85 years, into a 4-week exercise program. Participants will be allocated to one of the following groups using minimization, a type of randomization based on the lower extremity Fugl-Meyer score: 1) moderate intensity continuous training (MICT), that serves as the control, or 2) high-intensity interval training (HIIT). Exercise will be performed on a recumbent stepper. The Investigator will: Assess the preliminary efficacy of HIIT on aerobic fitness (Aim 1), cerebrovascular hemodynamics (Aim 2), and vascular function (Aim 3).

Current exercise recommendations for stroke use general exercise prescription principles for older adults and are not grounded on data generated from large, well-designed, randomized controlled trials in stroke. If aerobic exercise could be proven to reduce the number of "years of life lived with disability," it would offer a key strategy for: 1) minimizing dependence on caregiver support, 2) reducing overall healthcare costs, and 3) extending quality of life for individuals after stroke. This proposed trial will address an important gap in knowledge for both the scientific and clinical communities and provide essential data that will contribute to future exercise prescription recommendations focused on stroke.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes between the age of 20-85 years at time of consent
* Chronic ischemic or hemorrhagic stroke 6 months to 15 years at consent. People with stroke and newly diagnosed cardiovascular complications had >50% prevalence of recurrent stroke at 5 years. Index stroke or recurrent stroke on same side as index stroke will be allowed.
* Ability to walk over ground with assistive devices and no continuous physical assistance from another person to perform tests for gait speed and six-minute walk test
* Exercise continuously for minimum of 30 watts for 3 minutes on the recumbent stepper to demonstrate ability to perform the exercise test.
* No aerobic exercise contraindications or other safety/physical concerns during the submaximal exercise test.
* Able to communicate with investigators, follow 2-step command & correctly answer consent comprehension questions
* Currently participating in less than 150 minutes of physical activity/week assessed by the Rapid Assessment of Physical Activity
* Stable blood pressure & statin medication doses for 30 days prior to enrollment due to effects on vascular health/hemodynamics

Exclusion Criteria:

* Hospitalization for cardiac or pulmonary disease within past 3 months
* Implanted pacemaker or defibrillator limiting exercise performance
* Reported pain that limits or interferes with activities of daily living and physical activity/exercise
* Severe LE spasticity (Ashworth >2) due to inability to exercise
* Recent history (<3 months) of illicit drug or alcohol abuse or diagnosis of significant mental illness
* Major post-stroke depression (Patient Health Questionnaire, PHQ-9 ≥ 1084)
* Currently participating in physical therapy targeting lower extremity function or another interventional study that may influence study outcomes
* Other significant neurologic, orthopedic or peripheral vascular conditions that would limit exercise participation
* Oxygen-dependent chronic obstructive pulmonary disease
* Diagnosis of other neurological disease (Multiple Sclerosis, Alzheimer's disease, Parkinson's disease)
* Self report pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Oxygen uptake (VO2) | Baseline, 4 weeks
  Assessing change in oxygen uptake during a submaximal exercise test

SECONDARY OUTCOMES:
Middle cerebral artery velocity | Baseline, 4 weeks
  Assessing change in middle cerebral artery velocity response to an acute exercise bout
Middle cerebral artery velocity at rest | Baseline, 4 weeks
  Assessing change in middle cerebral artery velocity during a rest condition
Flow-mediated Dilation | Baseline, 4 weeks
  Endothelial vascular function
Pulse Wave Velocity | Baseline, 4 weeks
  Arterial stiffness

OTHER OUTCOMES:
6-Minute Walk Test (6MWT) | Baseline, 4 weeks
  Walking endurance using the 6MWT
10-Meter Walk Test | Baseline, 4 weeks
  Gait speed using the 10-Meter Walk Test
Cerebral Blood Flow | Baseline, 4 weeks
  Global and regional blood flow using MRI

CONTACTS AND LOCATIONS:
Overall Officials: Sandra A Billinger, PhD, Principal Investigator — KU Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Bartsch BL, Britton-Carpenter AJ, Engler A, Baldridge T, Moores A, Hazen EM, Montgomery RN, Billinger SA. Fitness After Stroke Trial (FAST): Protocol for a Preliminary Efficacy Study of Recumbent Stepper High-Intensity Interval Training. Res Sq [Preprint]. 2025 Dec 22:rs.3.rs-8264290. doi: 10.21203/rs.3.rs-8264290/v1. PMID 41510301